CLINICAL TRIAL: NCT06110676
Title: A Muti-center, Randomized, Double Blind, Positive Control Phase III Clinical Study to Evaluate the Efficacy and Safety of LZM012 in Moderate to Severe Chronic Plaque Psoriasis Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of LZM012
Acronym: Psoriasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LZM012-III
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LZM012 Q4W (Experimental): Patients receive 320mg of LZM012 treatment once every 4 weeks
  Interventions: Biological: LZM012
- LZM012 Q4W-Q8W (Experimental): Patients receive 320mg of LZM012 treatment once every 4 weeks till 12th week, then once evey 8 weeks
  Interventions: Biological: LZM012
- Active control (Active Comparator): Patients receive 300mg of secukinumab treatment once every 4 weeks
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: LZM012 — Recombinant anti-human IL-17A/F humanized monoclonal antibody injection
  Arms: LZM012 Q4W; LZM012 Q4W-Q8W
Biological: Secukinumab — Cosentyx
  Arms: Active control

SUMMARY:
This study is a muti-center, randomized, double blind, positive control phase III clinical study to evaluate the efficacy and safety of LZM012 in moderate to severe chronic plaque psoriasis patients

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 years at screening;
2. Patients with moderate to severe plaque psoriasis history with or without psoriatic arthritis for at least ≥6 months prior to baseline, and meet the following 3 criteria at screening and baseline:

   * PASI score ≥12
   * sPGA score ≥3
   * BSA ≥10%
3. Moderate to severe plaque psoriasis patients who are eligible for systemic therapy or phototherapy, defined as one of the following:

   * Insufficient efficacy after topical and/or phototherapy, photochemotherapy, and/or previous systemic therapy;
   * Intolerance to conventional therapy;
   * High SAE risk after conventional therapy;
   * Not suitable for conventional treatment due to comorbidities;
4. Patients meet the indications specified in the secukinumab label (i.e., adult patients with moderate to severe plaque psoriasis who meet the indications for systemic therapy or phototherapy) and had no contraindications as described in the secukinumab insert according to investigator's assessment;
5. Female patients must meet one of the following criteria:

   * Postmenopausal period. Menopause is defined as: 12 consecutive months of menopause in a woman over 40 years of age, excluding pregnancy and other conditions that may cause amenorrhea;
   * Permanent sterilization (e.g., tubal obstruction, hysterectomy, bilateral salpingectomy, etc.);
   * Women of childbearing potential who have no fertility or egg donation plans during treatment and for at least 6 months after the last trial drug treatment, and voluntarily use highly effective contraception (negative pregnancy test at screening and baseline); Male patients had no fertility or sperm donation plans during treatment and at least 6 months after the last trial drug treatment, and voluntarily took highly effective contraceptive measures;
6. Voluntarily participate in the study and sign an informed consent form (ICF) in writing, willing and able to comply with the study visit schedule and other requirements of the study protocol.

Exclusion Criteria:

1. Patients who are allergic to any component of the test drug, or who have had a severe allergic reaction to monoclonal antibodies, or who are judged by the investigator to be at risk of severe allergy to enter the study;
2. Patients with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, or drug-induced psoriasis at the time of screening;
3. Patients with progressive or uncontrolled systemic diseases such as kidney, liver, blood, gastrointestinal, endocrine, pulmonary, heart, neurological, psychiatric diseases, etc., who are not suitable to participate in this clinical trial according to the assessment of investigators due to the instability or possibility of development of the above diseases during the trial;
4. Patients with medical history, symptoms, signs or examination results suggested active tuberculosis, latent tuberculosis and inactive tuberculosis will be assessed by the investigators to participate in the trial or not;
5. Infectious diseases: a. patients with any serious infection within 1 month prior to baseline, defined as hospitalization due to infection or requiring intravenous anti-infective treatment; b. history of opportunistic infection or recurrent, chronic infection, which the investigator believes may lead participants to terminate the study; Opportunistic infections include infections caused by uncommon pathogens (e.g., Pneumocystis jirovecii, Cryptococcus, etc.) or unusually severe infections caused by common pathogens (e.g., cytomegalovirus, herpesvirus, etc.);
6. Patients with unstable cardiovascular and cerebrovascular diseases, defined as clinical deterioration phenomena (such as unstable angina, rapid atrial fibrillation, cerebral hemorrhage, acute cerebral infarction, etc.) within 3 months before screening, or hospitalization for cardiovascular and cerebrovascular diseases within 3 months before screening;
7. Patients with any history of active malignancy or malignancy in the 5 years prior to screening; except cured cancers (e.g. basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, localized low-risk prostate cancer, papillary thyroid cancer, etc.) and carcinoma in situ that has been radically resected (e.g. intraductal carcinoma in situ, carcinoma in situ of the cervix, etc.);
8. Patients with a history of lymphoproliferative disorders, including signs and symptoms of lymphoma or underlying lymphoproliferative disorders;
9. Patients with a history of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine) or history of illicit drug abuse in a year prior to screening;
10. Patients with inflammatory or autoimmune diseases other than psoriasis or psoriatic arthritis (e.g. inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, etc.);
11. Patients with a history of depression within one year prior to screening, or suicidal thoughts or any suicidal behavior assessed according to the Colombia-Suicide Severity Scale (C-SSRS) during the screening period or at baseline, patients who answered "yes" to any question on the C-SSRS questionnaire (questions 1~5), or patients who were clinically judged by the investigator to be at risk of suicide, will be excluded;
12. Patients who received topical anti-psoriasis therapy within 2 weeks prior to baseline, including:

    * topical therapeutic drugs/moisturizers/emollients/shampoos/shower gels containing moderate/potent/ultra-potent glucocorticoids, tretinoins, vitamin D3 derivatives, calcineurin inhibitors, α or β hydroxy acids, phosphodiesterase inhibitors, etc.;
    * Topical Chinese medicine/proprietary Chinese medicine with psoriasis therapeutic effect;
    * Drugs / moisturizer / emollient / shampoo / shower gel and other products containing urea, >3% salicylic acid, coal tar;
13. Patients received intra-articular corticosteroids 4 weeks or 5 half-lives (whichever is longer) before baseline;
14. Patients received physiotherapy (including psoralen and phototherapy/ photochemistry, tanning bed self-treatment, etc.) within 4 weeks before baseline;
15. Patients received non-biological systemic treatment of anti-psoriasis (including glucocorticoids, retinoids, cyclosporine, methotrexate, azathioprine, leflunomide, mycophenolate mofetil, tofacitinib, apremilast, traditional Chinese medicine/proprietary Chinese medicine, etc.) within 4 weeks before baseline
16. Patients received the following biologics or biosimilars prior to baseline:

    * Anti-tumor necrosis factor-α (TNF-α): etanercept < 28 days before baseline; Infliximab, golimumab, adalimumab, and Certolizumab Pegol < 90 days before baseline;
    * Anti-IL-12/IL-23 antibodies: ustekinumab < 6 months before baseline;
    * Anti-IL-23p19 antibodies: guselkumab < 90 days before baseline;
    * Rituximab or abatacept < 12 months before baseline;
17. Patients received anti-IL-17 antibody or anti-IL-17 receptor antibody therapy (including LZM012): e.g., secukinumab, ixekizumab, brodalumab, bimekizumab, or other test drugs against IL-17 antibodies or anti-IL-17 receptor antibodies;
18. Patients participated in clinical trials of any topical therapeutic agent (defined as have been administered) within 1 month before baseline;
19. Patients participated in a clinical trial (defined as have been administered) of any systemic therapeutic within 3 months before baseline or within 5 half-lives of the trial drug, whichever is longer;
20. Patients received a live vaccine (including live attenuated vaccine) within 3 months prior to baseline or plan to receive a live vaccine (including live attenuated vaccine) during the trial or within 6 months of the last trial drug administration; or plan to receive live shingles vaccine within 12 months of the last trial drug administration;
21. Lab test results meet any of the following conditions during screening period:

    * Blood routine: hemoglobin (HGB) <90g/L; Platelet count (PLT) < 100*109/L; Blood leukocytes (WBC) < 3*109/L; Absolute value (NEUT) of blood neutrophils< 1.5*109/L;
    * Liver function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeds the upper limit of normal value (ULN) by 3 times or total bilirubin exceeds 1.5 times the ULN;
    * Renal function: serum creatinine is greater than 1.5 times that of ULN;
    * Other abnormal laboratory test results, which may affect the subject's completion of the test or interfere with the test results as assessed by the investigator; Test could be repeated during the screening period for the false individual test results, or value near the limit, or inconclusive results, or according to the investigator's judgement. After re-test, subjects should not be randomized if the results still meet the above conditions;
22. Patients showed positive for hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV), or anti-syphilis spiral antibody (TP-Ab) [rapid plasma reagin ring card test (RPR) or toluidine red unheated serum test (TRUST) negative can be enrolled], or hepatitis B virus surface antigen (HBsAg);

    Under the condition of HBsAg negative, if:
    * Patients showed negative for all antigen antibodies of Hepatitis B, or positive for hepatitis B virus surface antibody (HBsAb)[with or without hepatitis B virus core antibody (HBcAb) positive], can be enrolled without hepatitis B virus DNA testing;
    * Patients showed HBsAb negative and HBcAb positive, HBV-DNA test is required. If HBV-DNA result showed negative or below the upper limit of normal, the patient can be enrolled;
23. Female subjects of childbearing potential tested positive for pregnancy during screening/baseline;
24. Lactating women;
25. Those considered by the investigator as inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
PASI100 response rate | At week 12
  The ratio of patients reached PASI100 (PASI100 response rate)

SECONDARY OUTCOMES:
PASI100 response rate | At week 52
  Compare the efficacy of LZM012 and Secukinumab
PASI 75 response rate | At week 4
  Compare the efficacy of LZM012 and Secukinumab
PASI 90 response rate | At week 12
  Compare the efficacy of LZM012 and Secukinumab
sPGA0/1 response rate | At week 12
  Compare the efficacy of LZM012 and Secukinumab

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China